CLINICAL TRIAL: NCT07142343
Title: An Open-Label, Single-Arm Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Pozelimab in Pediatric Patients 1 to 5 Years of Age With CD55-Deficient Protein-Losing Enteropathy (CHAPLE Disease)
Brief Title: A Study to Test the Safety of Pozelimab in Pediatric Participants 1 to 5 Years of Age With a Rare Disease Called CHAPLE (Complement Hyperactivation, Angiopathic Thrombosis, Protein-losing Enteropathy) Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PLE-2399
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: CHAPLE Disease
Keywords: CD55-deficient PLE (CHAPLE disease); CD55 loss-of-function mutation; Complement hyperactivation; Angiopathic thrombosis; Protein-losing enteropathy; Total Complement Hemolytic Activity Assay (CH50)
MeSH Terms: conditions — Protein-Losing Enteropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active CHAPLE (Experimental)
  Interventions: Drug: Pozelimab

INTERVENTIONS:
Drug: Pozelimab — Administered per the protocol
  Other Names: VEOPOZ

SUMMARY:
This study is researching a drug called pozelimab (called "study drug"). The main aim of this study is to monitor the safety and tolerability of the study drug.

The study is focused on young children 1 to 5 years of age, who have CHAPLE disease. CHAPLE is a very rare hereditary disease that can cause potentially life-threatening symptoms related to the stomach and intestines (gastrointestinal symptoms), and symptoms related to the heart and blood vessels (cardiovascular symptoms).

The study is also looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the study drug blocks Complement 5 (C5) in the body
* Whether the study drug changes the level of a substance called CH50 measured in the blood
* Whether the study drug changes the levels of albumin and other proteins
* Whether the body makes antibodies against study drug, which could make the study drug less effective or could lead to side effects

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical diagnosis of CD55-deficient CHAPLE disease as described in the protocol
2. Parent(s)/legal guardian(s) are willing and able to comply with participant's clinic visits and study-related procedures, including participant's completion of the full series of meningococcal vaccinations required per protocol.
3. Parent(s)/legal guardian(s) are willing to provide written informed consent
4. Participant has active CHAPLE disease as described in the protocol

Key Exclusion Criteria:

1. History of meningococcal infection
2. No documented meningococcal quadrivalent (serotype ACWY) vaccination prior to screening and participant's parent(s)/legal guardian(s) are unwilling for participant to undergo vaccination during the study as described in the protocol
3. No documented vaccination for Haemophilus influenzae and Streptococcus pneumoniae if applicable based on local practice or guidelines prior to screening as described in the protocol
4. Prior treatment with a complement inhibitor as described in the protocol
5. Presence of a concomitant disease that leads to hypoproteinemia or secondary intestinal lymphangiectasia as described in the protocol

Note: Other Protocol Defined Inclusion/ Exclusion Criteria Apply

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2026-03-06 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Event (TEAEs) | Through week 52
Severity of TEAEs | Through week 52

SECONDARY OUTCOMES:
Concentrations of total pozelimab | Through week 52
Concentrations of total C5 in serum | Through week 52
Absolute change from baseline of albumin concentration in serum | Through week 52
Percent change from baseline of albumin concentration in serum | Through week 52
Absolute change from baseline of total protein | Through week 52
Percent change from baseline of total protein | Through week 52
Absolute change from baseline of total Immunoglobulin G (IgG) | Through week 52
Percent change from baseline of total IgG | Through week 52
Incidence of Anti-Drug Antibody (ADA) to pozelimab over time | Through week 52
Titer of ADA to pozelimab over time | Through week 52
Change from baseline of total complement activity CH50 over time | Through week 52
Percent change from baseline of CH50 over time | Through week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/